CLINICAL TRIAL: NCT02977559
Title: A Comparative Randomized Prospective Study Between the New Laryngeal Tube Suction-Disposable and the Ambu AuraGain in Pediatric Patients
Brief Title: A Study Between the Laryngeal Tube Suction-Disposable and the Ambu AuraGain in Pediatric Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, LUIS.GAITINI, medical doctor, Bnai Zion Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BnaiZionMC-16-LG-012
Record Dates: First submitted 2016-11-28; First posted 2016-11-30 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Adverse Anesthesia Outcome
Keywords: Laryngeal Tube Suction Ambu AuraGain Leak Pressure

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laryngeal Tube Suction Disposable (Experimental): Laryngeal Tube Suction Disposable for ventilation
  Interventions: Device: Laryngeal Tube Suction Disposable
- Laryngeal Mask Airway AuraGain (Experimental): Laryngeal Mask Airway AuraGain for oxygenation and ventilation
  Interventions: Device: Laryngeal Mask Airway AuraGain

INTERVENTIONS:
Device: Laryngeal Tube Suction Disposable — Device for ventilation
  Arms: Laryngeal Tube Suction Disposable
Device: Laryngeal Mask Airway AuraGain — Ventilation device
  Arms: Laryngeal Mask Airway AuraGain

SUMMARY:
The study compared the Laryngeal Tube Suction Disposable (LTS-D) with the Disposable Laryngeal Mask Ambu® AuraGain™ (DLMA AG) during general anesthesia in pediatric patients.

The investigators hypothesized that the LTS-D and the DLMA AG performed similarly during mechanical ventilation despite differences in their structural design.

DETAILED DESCRIPTION:
The Laryngeal Tube Suction-Disposable (LTS-D, (VBM Medizintechnik GmbH, Sulz, Germany), is a second generation single-use supraglottic airway devices (SADs) with gastric access, for airway management in spontaneously and mechanically ventilated patients undergoing general anesthesia.

The AuraGain is a second generation laryngeal mask, satisfying airway management needs by integrating gastric access and ventilation capability in an anatomically curved single-use device that facilitates rapid establishment of a safe airway.

The two devices have now pediatric sizes.

To date, there is no published data comparing the LTS-D and the DLMA AG during mechanical ventilation in pediatric patients. The investigators hypothesized that the LTS-D and the DLMA AG perform similarly during mechanical ventilation despite differences in their structural design.

The chief aim of this prospective randomized study was to compare the LTS-D and the DLMA AG with respect to:

1. time to achieve an effective airway,
2. ease of insertion,
3. need for interventions to achieve an effective airway,
4. cuff seal (leak) pressure at an intracuff pressure of 60 cm H2O,
5. ventilatory variables during mechanical ventilation,
6. fiberoptic score,
7. gastric tube insertion and
8. adverse perioperative events.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients, American Society of Anesthesiologist (ASA) physical status I and II weighing 30 to 10 kg, posted for abdominal surgery under general anesthesia.

Exclusion Criteria:

* Infants with active respiratory tract infection anticipated and known difficult airway, lung disease requiring high positive end expiratory pressure, and active gastrointestinal reflux will be excluded.

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2017-03; Primary Completion 2017-04 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Leak pressure measure in cm H2O | 60 seconds

SECONDARY OUTCOMES:
Time to insertion a device in seconds | 60 seconds

IPD SHARING:
Plan to Share IPD: Yes